CLINICAL TRIAL: NCT04301557
Title: PD1 Antibody Toripalimab and Chemoradiotherapy for dMMR/MSI-H Locally Advanced Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuan-hong Gao, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-177-01
Record Dates: First submitted 2020-02-23; First posted 2020-03-10 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: DMMR Colorectal Cancer; MSI-H Colorectal Cancer; Locally Advanced Colorectal Cancer
Keywords: DMMR Colorectal Cancer; MSI-H Colorectal Cancer; Locally Advanced Colorectal Cancer
MeSH Terms: interventions — spartalizumab; toripalimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD1 Antibody and Chemoradiotherapy for dMMR/MSI-H LACRC (Experimental): Induction regimen: Capeox+PD1 antibody for 1 cycle, Concurrent chemoradiotherapy regimen: Capeox+PD1 antibody for 2 cycles and concurrent , Interval regimen: Capeox+PD1 antibody for 1 cycle, TME surgery or watch and wait for cCR patients Adjuvant regimen: Capeox+PD1 antibody for 2 cycles, Capecitabine+PD1 antibody for 2 cycles
  Interventions: Drug: PD-1 Antibody; Drug: Oxaliplatin; Drug: Capecitabine; Radiation: External beam radiotherapy; Procedure: Total mesorectal excision

INTERVENTIONS:
Drug: PD-1 Antibody — PD-1 antibody 240mg,I.V,D1,repeat every 3 weeks, Four cycles in the neoadjuvant treatment, and four cycles in the adjuvant treatment,
  Other Names: Toripalimab
Drug: Oxaliplatin — Oxiliplatin 130mg/m^2 (100mg/m^2 during radiotherapy),I.V,D1,repeat every 3 weeks, Four cycles in the neoadjuvant treatment in Capeox regimen, and two cycles in the adjuvant treatment in Capeox regimen
Drug: Capecitabine — Capecitabine 1000mg/m^2,Bid,P.O,D1-D14,repeat every 3 weeks, Four cycles in the neoadjuvant treatment in Capeox regimen, and two cycles in the adjuvant treatment in Capeox regimen, and two cycles in adjuvant treatment in Capecitabine regimen
Radiation: External beam radiotherapy — Neoadjuvant radiotherapy, 50Gy/25Fractions to the GTV, 45Gy/25Fractions to the CTV
Procedure: Total mesorectal excision — Total mesorectal excision

SUMMARY:
PD1 antibody is now recommended for dMMR/MSI-H metastatic colorectal cancer patients as second line. Chemoradiotherapy is standand treatment for locally advanced rectal cancer and is also recommended as an alternative choice for unresectable locally advanced colon cancer. Thus, this study will investigate the efficacy and toxicity of combination strategy using PD1 antibody and chemoradiotherapy for dMMR/MSI-H locally advnaced colorectal cancer patients.

DETAILED DESCRIPTION:
PD1 antibody is recommended for dMMR/MSI-H metastatic colorectal cancer patients as second line. Chemoradiotherapy is standand treatment for locally advanced rectal cancer and is also recommended as an alternative choice for unresectable locally advanced colon cancer. Thus, this phase II, single arm study will investigate the efficacy and toxicity of combination strategy using PD1 antibody and chemoradiotherapy for dMMR/MSI-H locally advnaced colorectal cancer patients, which is expected to yield higher tumor regressiona with tolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of colorectal adenocarcinoma;
2. Biopsy tissues with IHC indicates deficient mismatch repair(dMMR),that is,the loss of at least one of the four proteins ,MSH1,MSH2,MSH6,PMS2;or gene detection implies MSI-H;
3. Clinical stage for rectal cancer patients is cT3-4N0M0 or cTxN+M0;clinical stage of colon cancer should meet the following criteria (any one is sufficient): a)Tumor penetrates the whole wall and adherents to other organs or structures around(T4b).Tumor cannot reach R0 resection by imaging assessment; b)The intestinal lymph nodes involved are closely adjacent to large abdominal vessels. Lymph nodes dissection is not feasible by imaging assessment; c)Surgeons assess it is hard to achieve R0 resection after surgical exploration; d)Surgeons assess tumor is extensive multiviseral resection is needed, which is expected to damage the organs and seriously affect the quality of life after operation;
4. Preoperative staging methods: all patients need to accept digital rectal examination(DRE).Patients with rectal cancer undergo high-resolution MRI±ultrasound colonoscopy/transrectal ultrasound for preoperative staging. Perienteric lymph nodes with short diameter ≥10mm or the shape of lymph nodes and its MRI characteristics are consistent with typical lymph node metastasis. If endoscopic ultrasonography is used in combination, and there is a contradiction between staging methods, the data should be submitted to the evaluation team of our center for the accurate staging;
5. No symptoms of ileus; or ileus is alleviated after proximal colostomy.

Previous treatment:

1. No surgery except preventative stoma;
2. No chemotherapy or radiotherapy;
3. No biotherapy (e.g.monoclonal antibodies), immunotherapy (e.g.anti-PD-1 antibody,anti-PD-L1 antibody,anti-PD-L2 antibody or CTLA-4 antibody),or other clinical trials agents;
4. No limit to previous endocrine therapy.

Patient characteristics:

1. Age between 18 and 72 years;
2. ECOG performance status of 0 or 1;
3. Life expectancy: more than 2 years;
4. Hematopoietic: WBC>3×109/L;PLT>80×109/L; Hb>90g/L;
5. Hepatic: ALT and AST<2 times upper limit of normal (ULN); bilirubin<1.5 times ULN;
6. Renal: creatinine <1.5 times ULN or creatinine clearance ≥ 60 mL/min.

Exclusion Criteria:

All patients enrolled cannot have any of the following situation:

1. Arrhythmias require antiarrhythmic therapy (with the exception of β-blockers or digoxin), symptomatic coronary artery disease or local myocardial ischemia (myocardial infarction within the past 6 months) or congestive heart failure exceeding NYHA II;
2. Severe hypertension with poor drug control;
3. A known history of testing positive for HIV or chronic hepatitis B or C (high copy virus DNA) at active stage;
4. Patients with active tuberculosis (TB) are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening;
5. Other active severe clinical infections (NCI-CTC5.0);
6. Apparent distant metastasis away from the pelvic before surgery;
7. Cachexia, organ function decompensation;
8. Previous pelvic or abdominal radiotherapy;
9. Multiple primary colorectal cancers;
10. Epilepsy require medical treatment (such as steroid or antiepileptic therapy);
11. Other malignancy within the past 5 years with the exception of effectively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin;
12. Drug abuse and medical, psychological or social factors that may interfere with patients' participation in the study or affect the evaluation of the study;
13. Patients have any active autoimmune diseases or a history of autoimmune diseases(including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism and decreased thyroid function; patients with vitiligo or with complete remission of asthma in childhood and without any intervention in adulthood may be included; patients with asthma requiring bronchodilators intervention are not included.
14. Received any anti-infection vaccine (e.g. influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before enrollment;
15. Complications require long-term treatment with immunosuppressive drugs, or requiring systemic or local use of immunosuppressive corticosteroids(>10mg/day prednisone or other therapeutic hormones);
16. Known or suspected allergy to the study drugs or to any drugs related to this trial;
17. Any unstable condition or which endangers the patients' safety and compliance;
18. Pregnant or breast-feeding women who are fertile without effective contraception;
19. Refuse to sign the informed consent.

Exit Criteria:

1. Patients withdraw the informed consent and ask for quit;
2. Poor compliance;
3. Disease progression during treatment;
4. Serious adverse events or serious adverse reactions (SAE) occurred during the study;
5. Any delay of treatment for more than two weeks (including two weeks) (referring to the delay of all drugs in the medication plan) shall be discussed by the researchers whether to quit.

Cessation Criteria:

Study suspension refers to the cessation of the whole study before the end of the program. The main purpose of this action is to protect the rights and interests of the subjects, ensure the quality of the study, and avoid unnecessary economic losses. The whole study will be stopped for the following reasons:

1. Researchers find serious safety issues;
2. Efficacy is poor that there is no need to continue the study;
3. Severe mistakes in the scheme design or important deviations in the implementation process;
4. Funds or management problems;
5. The administrative department decide to cancel the study. A complete suspension of research is either temporary or permanent. When discontinued, all study records shall be retained for future reference.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2024-04-22 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response(pCR) | 1 week after surgery
  According to pathological response to assess the efficiency of treatment

SECONDARY OUTCOMES:
Acute toxicities | Up to 3 months after adjuvant treatment
  Acute toxicities according to CTCAE5.0
Tumor regression grade | 1 week after surgery
  Tumor regression grade
R0 resection rate | 1 week after surgery
  R0 resection rate
Surgical Complication | Surgery scheduled 6-8 weeks after the end of neoadjuvant treatment
  Surgical Complication
Local recurrence | From date of randomization until the date of local recurrence, assessed up to 10 years
  Local recurrence
Distant metastasis | From date of randomization until the date of death of distant metastasis, assessed up to 10 years
  Distant metastasis
3 year disease free survival | From date of randomization until the date of disease recurrence, assessed up to 3 years
  3 year disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corrigendum to "Neoadjuvant 5-FU or Capecitabine Plus Radiation With or Without Oxaliplatin in Rectal Cancer Patients: A Phase III Randomized Clinical Trial". J Natl Cancer Inst. 2018 Jul 1;110(7):794. doi: 10.1093/jnci/djy096. No abstract available. PMID 29800481
- [Background] Croner RS, Merkel S, Papadopoulos T, Schellerer V, Hohenberger W, Goehl J. Multivisceral resection for colon carcinoma. Dis Colon Rectum. 2009 Aug;52(8):1381-6. doi: 10.1007/DCR.0b013e3181ab580b. PMID 19617748
- [Background] Lehnert T, Methner M, Pollok A, Schaible A, Hinz U, Herfarth C. Multivisceral resection for locally advanced primary colon and rectal cancer: an analysis of prognostic factors in 201 patients. Ann Surg. 2002 Feb;235(2):217-25. doi: 10.1097/00000658-200202000-00009. PMID 11807361
- [Background] Eldar S, Kemeny MM, Terz JJ. Extended resections for carcinoma of the colon and rectum. Surg Gynecol Obstet. 1985 Oct;161(4):319-22. PMID 4049200
- [Background] Chang H, Yu X, Xiao WW, Wang QX, Zhou WH, Zeng ZF, Ding PR, Li LR, Gao YH. Neoadjuvant chemoradiotherapy followed by surgery in patients with unresectable locally advanced colon cancer: a prospective observational study. Onco Targets Ther. 2018 Jan 17;11:409-418. doi: 10.2147/OTT.S150367. eCollection 2018. PMID 29398921
- [Background] Curley SA, Carlson GW, Shumate CR, Wishnow KI, Ames FC. Extended resection for locally advanced colorectal carcinoma. Am J Surg. 1992 Jun;163(6):553-9. doi: 10.1016/0002-9610(92)90554-5. PMID 1595834
- [Background] Xin Yu, WeiWei Xiao, Rong Zhang, LuNing Zhang, Bo Qiu, ZhiFan Zeng, Pei-Rong Ding, Zhi-zhong Pan, Li-ren LI, Yuan-Hong Gao. A pilot study of neoadjuvant chemoradiotherapy for unresectable locally advanced adherent colon cancer: Assessing local tumor response. JCO. 2016; 34（4S）: 727.
- [Background] Qiu B, Ding PR, Cai L, Xiao WW, Zeng ZF, Chen G, Lu ZH, Li LR, Wu XJ, Mirimanoff RO, Pan ZZ, Xu RH, Gao YH. Outcomes of preoperative chemoradiotherapy followed by surgery in patients with unresectable locally advanced sigmoid colon cancer. Chin J Cancer. 2016 Jul 7;35(1):65. doi: 10.1186/s40880-016-0126-y. PMID 27389519
- [Background] Cukier M, Smith AJ, Milot L, Chu W, Chung H, Fenech D, Herschorn S, Ko Y, Rowsell C, Soliman H, Ung YC, Wong CS. Neoadjuvant chemoradiotherapy and multivisceral resection for primary locally advanced adherent colon cancer: a single institution experience. Eur J Surg Oncol. 2012 Aug;38(8):677-82. doi: 10.1016/j.ejso.2012.05.001. Epub 2012 May 24. PMID 22632848
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Lemery S, Keegan P, Pazdur R. First FDA Approval Agnostic of Cancer Site - When a Biomarker Defines the Indication. N Engl J Med. 2017 Oct 12;377(15):1409-1412. doi: 10.1056/NEJMp1709968. No abstract available. PMID 29020592
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Diaz LA Jr, Le DT. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Nov 12;373(20):1979. doi: 10.1056/NEJMc1510353. No abstract available. PMID 26559582